CLINICAL TRIAL: NCT04844190
Title: Use of Endoscopic Functional Lumen Imaging Probe (EndoFLIP) and Antroduodenal Manometry (ADM) in Predicting Clinical Response to Gastric Peroral Endoscopic Myotomy (G-POEM): A Pilot Study
Brief Title: Use of EndoFLIP and Manometry Prior to G-POEM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to complete study procedures due to staffing issues.
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00213007
Record Dates: First submitted 2021-03-11; First posted 2021-04-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Gastroparesis
Keywords: G-POEM; High Resolution Manometry; Endoscopic Functional Lumen Imaging Probe
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Intervention Model Description: Prospective Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Addition of ADM and EndoFLIP to pre-G-POEM evaluation (Experimental): During the preoperative upper endoscopy, the EndoFLIP catheter is inserted through the mouth with endoscopic guidance and placed through the gastric pylorus. Once deployed, water is sequentially added at set volumes to a balloon that can be used to measure pyloric diameter, cross-sectional area, pressure, and distensibility at set volumes of 30, 40, and 50 mL for at least five seconds. We will record this data for each patient. The EndoFLIP catheter will then be removed. Subsequently, a high resolution ADM catheter will be inserted through the nose and placed through the pylorus to measure baseline intragastric, transpyloric, and intraduodenal pressures. The patient will be observed for up to four hours to assess a migrating motor complex (MMC). After the MMC is observed, the patient will be given a meal and observed for meal response with the manometry catheter. The meal will be water and two pieces of toast/bread. Following the meal, the catheter will be removed.
  Interventions: Diagnostic Test: EndoFLIP; Diagnostic Test: Antroduodenal Manometry

INTERVENTIONS:
Diagnostic Test: EndoFLIP — During pre-G-POEM upper endoscopy, an EndoLIP catheter will be inserted through the patient's mouth into the stomach and across the pylorus. Once results of EndoFLIP are obtained, the catheter will be removed (5 minutes).
Diagnostic Test: Antroduodenal Manometry — Following removal the EndoFLIP catheter, a manometry catheter will then be placed through the nose and advanced across the pylorus. Once catheter positioning is confirmed on endoscopy, the endoscope will be withdrawn. The manometry catheter will be taped to the nose and sedation stopped. The patient will be brought to the recovery area where they will wake-up with the catheter in place. In a private recovery room, the patient will have the catheter in place (no positioning or movement restrictions). When pyloric spasms are documented (0.5-4 hours), they will be given a standard small meal (water, toast/bread). Once motility is assessed with eating, the manometry catheter will be removed.

SUMMARY:
The purpose of this study is to assess physiologic response of therapy in patients with refractory gastroparesis undergoing Gastric per-oral endoscopic myotomy (G-POEM) using endoscopic functional lumen imaging probe (EndoFLIP) and antroduodenal manometry (ADM). Refractory gastroparesis will be defined as having delayed gastric emptying at four hours (>10% retention of stomach contents) on gastric scintigraphy and persistent symptoms despite treatment with dietary modification or prokinetic medications. We hypothesize that EndoFLIP and high resolution ADM will provide an individualized pyloric functional profile in gastroparesis patients that can more accurately predict clinical response to G-POEM.

DETAILED DESCRIPTION:
Gastroparesis is defined as an objective delay in gastric emptying in the absence of mechanical obstruction with corresponding cardinal symptoms of postprandial fullness, early satiety, nausea, vomiting, bloating, and abdominal pain. Gastroparesis-related hospitalizations have increased by 158% in recent years as healthcare costs associated with gastroparesis have similarly risen exponentially by 1026% from 1997 to 2013.

Medical management of gastroparesis, primarily comprised of dietary and prokinetic therapy, is limited in effectiveness, tolerability, and durability, in part because the pathophysiologic mechanisms underlying gastroparesis are varied and multifactorial, including pyloric dysfunction, impaired fundic accommodation, vagal injury or neuropathy, gastric pacemaker dysrhythmias, hypocontractility, and aberrant gastric feedback. Pyloric dysfunction in particular, characterized by increased tone or pylorospasm, offers the potential for targeted endoscopic therapy in a subset of patients.

Gastric peroral endoscopic myotomy (G-POEM) has recently emerged as a feasible and safe treatment for severe refractory gastroparesis. Initially described in 2013, G-POEM is a minimally invasive technique that consists of creating a submucosal tunnel extending to the pylorus, dissecting circular and oblique muscle layers, and closing the tunnel with endoscopic clips. The first systematic review of early outcomes of G-POEM across 10 studies and 292 patients revealed 100% technical success, symptomatic improvement in 84%, and an adverse event rate of 6.8%.

However, a nuanced approach to appropriate patient selection for G-POEM, based on individual physiologic characteristics, is still lacking. The endoscopic functional lumen imaging probe (EndoFLIP; Crospon Inc., Galway, Ireland), previously well-described in assessing the lower esophageal sphincter in esophageal motility disorders, has been recently proposed as an adjunctive technology for evaluating pyloric sphincter compliance and distensibility. Few studies have investigated the efficacy of pyloric EndoFLIP in gastroparesis. Gourcerol et al. reported that gastroparesis patients have lower pyloric compliance compared to healthy volunteers, which also correlated with longer gastric emptying half times and reduced quality of life scores. A second pilot study of 20 gastroparesis patients who underwent pre- and post-myotomy EndoFLIP revealed that a distensibility index of <9.2 mm2/mmHg was associated with G-POEM clinical efficacy, however the study was limited by a short follow-up time of three months.

Antroduodenal manometry (ADM) has been the gold standard of assessing pyloric function and early studies revealed elevated pyloric pressures in greater than 50% of diabetics with gastroparesis. Recent data also shows a significant correlation between manometric and EndoFLIP pressures, though to date, no studies have utilized ADM in evaluating the efficacy of G-POEM. While conventional ADM was previously felt to be technically challenging and limited in availability, the advancement of high resolution manometry presents a unique opportunity for complementary assessment of not only pyloric pressures, but also antroduodenal pressure gradients.

We propose that the use of both EndoFLIP and high resolution ADM will provide an individualized pyloric functional profile in gastroparesis patients that can more accurately predict clinical response to G-POEM. As one of only few nationwide centers performing G-POEM, Northwestern Medicine has one of the highest volumes of this novel endoscopic treatment, having successfully completed 40 procedures within the last year.

Adult patients with refractory gastroparesis will be enrolled in this prospective study. Refractory gastroparesis will be defined as having delayed gastric emptying at four hours (>10% retention) on gastric scintigraphy and persistent symptoms despite treatment with dietary modification or prokinetic medications. Preoperatively, patients will complete validated symptom and quality of life questionnaires, including the Gastroparesis Cardinal Symptom Index (GCSI), Patient Assessment of Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM), and Short Form 36 (SF-36). Patients will also complete an upper gastrointestinal series (UGIS) to evaluate the anatomy of the stomach. Patients will then undergo study protocol including G-POEM. Patients will be required to follow-up at one, three, and six months in clinic or via telephone visit following G-POEM to evaluate clinical response, identify any adverse events related to the procedure, and complete symptom and quality of life questionnaires. Per standard of care, repeat gastric scintigraphy will be obtained at three months following G-POEM and will be shared with study staff. The endpoints for this study following completion of 20 G-POEM procedures are:

Primary endpoint: To assess the predictive value of EndoFLIP for clinical response to G-POEM in patients with refractory gastroparesis. Clinical response will be defined as a decrease of 1 point in the average total GCSI score, comprised of a 6-point scoring system with 9 questions from 3 cardinal subscales, with more than 25% decrease in at least 2 of 3 subscales (nausea/vomiting, postprandial fullness/early satiety, and bloating).

Secondary endpoints: To assess the predictive value of high resolution ADM for clinical response to G-POEM in patients with refractory gastroparesis. Mean intragastric-intraduodenal pressure gradients averaged over one minute within a deflated stomach during upper endoscopy will be calculated for each patient.

To evaluate correlations between EndoFLIP pressure and distensibility and ADM transpyloric pressure and intragastric-intraduodenal pressure gradient.

Additional secondary endpoints include assessment of quality of life, objective gastric emptying, UGIS results, technical success of G-POEM, procedure time, and adverse event rate.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18+ diagnosed with refractory gastroparesis as defined earlier in this document, no age limit
* Patients already consented to undergo G-POEM

Exclusion Criteria:

* Patients who are pregnant(at Northwestern, all female patients have urine pregnancy tests on day of endoscopy), vulnerable populations such as prisoners,
* Life expectancy < 1 year based on concurrent comorbidities based on study team assessment,
* Coagulopathy with INR > 1.5 that cannot be reversed,
* Thrombocytopenia with platelets < 50,000 that cannot be corrected with blood products,
* Unable to safely undergo elective endoscopy due to current comorbidities, and inability to pass standard endoscope.
* Patients with history of gastric surgery and
* Active narcotic use at time of G-POEM evaluation within four weeks. Tobacco use is not an exclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Predictive Value of EndoFLIP | 24 months
  To assess the predictive value of EndoFLIP for clinical response to G-POEM in patients with refractory gastroparesis. We hypothesize that patients with lower pyloric distensibility (measured in mm2/mmHg) will be predictive of clinical response to G-POEM.
Predictive Value of ADM | 24 months
  To assess the predictive value of high resolution ADM for clinical response to G-POEM in patients with refractory gastroparesis. We hypothesize that patients with a large, positive pressure gradient will be predictive of clinical response to G-POEM.

SECONDARY OUTCOMES:
EndoFLIP data correlation | 24 months
  To evaluate correlations between EndoFLIP pressure and distensibility and ADM transpyloric pressure and intragastric-intraduodenal pressure gradient. We hypothesize that there will be significant negative correlation between pyloric distensibility and the intragastric-intraduodenal pressure gradient.
Quality of Life outcome of G-POEM | 36 months
  To further assess quality of life changes following G-POEM using Patient Assessment of Upper GI Symptoms (PAGI-SYM) questionnaire
Quality of Life outcome assessed by SF-36 QOL survey questionnaire | 36 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 36 months
  To monitor for adverse associated with G-POEM
Gastric-Emptying Characteristics | 36 months
  To assess changes in Gastric-Emptying Studies pre-procedure and post-procedure in percentage emptied at 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Camilleri M, Parkman HP, Shafi MA, Abell TL, Gerson L; American College of Gastroenterology. Clinical guideline: management of gastroparesis. Am J Gastroenterol. 2013 Jan;108(1):18-37; quiz 38. doi: 10.1038/ajg.2012.373. Epub 2012 Nov 13. PMID 23147521
- [Result] Wang YR, Fisher RS, Parkman HP. Gastroparesis-related hospitalizations in the United States: trends, characteristics, and outcomes, 1995-2004. Am J Gastroenterol. 2008 Feb;103(2):313-22. doi: 10.1111/j.1572-0241.2007.01658.x. Epub 2007 Nov 28. PMID 18047541
- [Result] Wadhwa V, Mehta D, Jobanputra Y, Lopez R, Thota PN, Sanaka MR. Healthcare utilization and costs associated with gastroparesis. World J Gastroenterol. 2017 Jun 28;23(24):4428-4436. doi: 10.3748/wjg.v23.i24.4428. PMID 28706426
- [Result] Camilleri M, Bharucha AE, Farrugia G. Epidemiology, mechanisms, and management of diabetic gastroparesis. Clin Gastroenterol Hepatol. 2011 Jan;9(1):5-12; quiz e7. doi: 10.1016/j.cgh.2010.09.022. Epub 2010 Oct 15. PMID 20951838
- [Result] Clarke JO, Snape WJ Jr. Pyloric sphincter therapy: botulinum toxin, stents, and pyloromyotomy. Gastroenterol Clin North Am. 2015 Mar;44(1):127-36. doi: 10.1016/j.gtc.2014.11.010. Epub 2015 Jan 13. PMID 25667028
- [Result] Khashab MA, Stein E, Clarke JO, Saxena P, Kumbhari V, Chander Roland B, Kalloo AN, Stavropoulos S, Pasricha P, Inoue H. Gastric peroral endoscopic myotomy for refractory gastroparesis: first human endoscopic pyloromyotomy (with video). Gastrointest Endosc. 2013 Nov;78(5):764-8. doi: 10.1016/j.gie.2013.07.019. No abstract available. PMID 24120337
- [Result] Spadaccini M, Maselli R, Chandrasekar VT, Anderloni A, Carrara S, Galtieri PA, Di Leo M, Fugazza A, Pellegatta G, Colombo M, Palma R, Hassan C, Sethi A, Khashab MA, Sharma P, Repici A. Gastric peroral endoscopic pyloromyotomy for refractory gastroparesis: a systematic review of early outcomes with pooled analysis. Gastrointest Endosc. 2020 Apr;91(4):746-752.e5. doi: 10.1016/j.gie.2019.11.039. Epub 2019 Dec 3. PMID 31809720
- [Result] Gourcerol G, Tissier F, Melchior C, Touchais JY, Huet E, Prevost G, Leroi AM, Ducrotte P. Impaired fasting pyloric compliance in gastroparesis and the therapeutic response to pyloric dilatation. Aliment Pharmacol Ther. 2015 Feb;41(4):360-7. doi: 10.1111/apt.13053. Epub 2014 Dec 19. PMID 25523288
- [Result] Jacques J, Pagnon L, Hure F, Legros R, Crepin S, Fauchais AL, Palat S, Ducrotte P, Marin B, Fontaine S, Boubaddi NE, Clement MP, Sautereau D, Loustaud-Ratti V, Gourcerol G, Monteil J. Peroral endoscopic pyloromyotomy is efficacious and safe for refractory gastroparesis: prospective trial with assessment of pyloric function. Endoscopy. 2019 Jan;51(1):40-49. doi: 10.1055/a-0628-6639. Epub 2018 Jun 12. PMID 29895073
- [Result] Mearin F, Camilleri M, Malagelada JR. Pyloric dysfunction in diabetics with recurrent nausea and vomiting. Gastroenterology. 1986 Jun;90(6):1919-25. doi: 10.1016/0016-5085(86)90262-3. PMID 3699409
- [Result] Snape WJ, Lin MS, Agarwal N, Shaw RE. Evaluation of the pylorus with concurrent intraluminal pressure and EndoFLIP in patients with nausea and vomiting. Neurogastroenterol Motil. 2016 May;28(5):758-64. doi: 10.1111/nmo.12772. Epub 2016 Jan 27. PMID 26813266
- [Result] Desipio J, Friedenberg FK, Korimilli A, Richter JE, Parkman HP, Fisher RS. High-resolution solid-state manometry of the antropyloroduodenal region. Neurogastroenterol Motil. 2007 Mar;19(3):188-95. doi: 10.1111/j.1365-2982.2006.00866.x. PMID 17300288
- [Result] Revicki DA, Rentz AM, Dubois D, Kahrilas P, Stanghellini V, Talley NJ, Tack J. Development and validation of a patient-assessed gastroparesis symptom severity measure: the Gastroparesis Cardinal Symptom Index. Aliment Pharmacol Ther. 2003 Jul 1;18(1):141-50. doi: 10.1046/j.1365-2036.2003.01612.x. PMID 12848636
- [Result] Rentz AM, Kahrilas P, Stanghellini V, Tack J, Talley NJ, de la Loge C, Trudeau E, Dubois D, Revicki DA. Development and psychometric evaluation of the patient assessment of upper gastrointestinal symptom severity index (PAGI-SYM) in patients with upper gastrointestinal disorders. Qual Life Res. 2004 Dec;13(10):1737-49. doi: 10.1007/s11136-004-9567-x. PMID 15651544
- [Result] Mekaroonkamol P, Patel V, Shah R, Li B, Luo H, Shen S, Chen H, Shahnavaz N, Dacha S, Keilin S, Willingham FF, Christie J, Cai Q. Association between duration or etiology of gastroparesis and clinical response after gastric per-oral endoscopic pyloromyotomy. Gastrointest Endosc. 2019 May;89(5):969-976. doi: 10.1016/j.gie.2018.12.023. Epub 2019 Jan 14. PMID 30653937